CLINICAL TRIAL: NCT05227755
Title: High-protein Oral Supplement Improves Normalized Protein Catabolic Rate and Inflammation Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB202101921; OCR41389 (Other: UF OnCore)
Record Dates: First submitted 2021-12-21; First posted 2022-02-07 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Renal Failure; Chronic Kidney Disease Requiring Chronic Dialysis
MeSH Terms: conditions — Renal Insufficiency | interventions — Soybean Proteins

STUDY DESIGN:
Intervention Model Description: This is a 12-week interventional, double-blind randomized controlled crossover clinical trial designed to evaluate the impact of whey (control) and soy (intervention) protein isolate oral supplements on protein status and inflammation markers.
Who Masked: Participant, Investigator
Masking Description: A third party vendor will provide the coded samples. The vendor will only reveal the actual products once the study has ended and analysis has occurred.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whey protein isolate (Active Comparator): Participants will receive 120 mls of whey protein isolate (total of 20 g protein) to consume 3x/week after dialysis treatment for 4 weeks.
  Interventions: Dietary Supplement: Whey protein isolate
- Soy protein isolate (Experimental): Participants will receive 120 mls of soy protein isolate (total of 20 g protein) to consume 3x/week after dialysis treatment for 4 weeks.
  Interventions: Dietary Supplement: Soy protein isolate

INTERVENTIONS:
Dietary Supplement: Soy protein isolate — Participants will receive 120 mls of soy protein isolate (total of 20 g protein) to consume 3x/week after dialysis treatment for 4 weeks.
  Arms: Soy protein isolate
Dietary Supplement: Whey protein isolate — Participants will receive 120 mls of whey protein isolate (total of 20 g protein) to consume 3x/week after dialysis treatment for 4 weeks.
  Arms: Whey protein isolate

SUMMARY:
The investigators propose to determine the impact of high-protein beverages on protein status and inflammation markers among CKD patients undergoing hemodialysis. A 12-week double-blind randomized cross-over trial will be used in which participants (n=22) will consume a 4-ounce high protein supplement with either whey (20 g total protein) or soy (20 g total protein). Outcomes of interest include serum urea nitrogen and inflammation markers (CRP and IL-6). The findings will contribute to the knowledge gap regarding the effect of different protein types in CKD populations which can be translated to the development of affordable supplements to prevent malnutrition in adults with non-communicable diseases.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* diagnosed with stage 5 CKD for at least 3 months prior to the starting date of the trial
* 3 sessions of hemodialysis per week for at least three months prior to the starting date of the trial
* All participants have the ability to provide signed informed consent
* have not been newly diagnosed
* not present with symptomatic infection of COVID-19
* have no dietary restriction
* no food allergies
* no chewing/swallowing difficulties

Exclusion Criteria:

* CKD patient stages 1-4.
* CKD patient undergoing peritoneal hemodialysis.
* In isolation due to COVID-19 or other infectious disease
* Adult pregnant and/or lactating for the duration of the study.
* Any other renal disease autoimmune or otherwise.
* Use of other IP within 3 months prior of the eligibility screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-08-05 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-11-21 (Actual)

PRIMARY OUTCOMES:
C-reactive protein | Up to 12 weeks of the study
  Collection of serum C-reactive protein to identify a change from pre-post to analyze the effect protein isolates had on inflammation markers.
IL-6 | Up to 12 weeks of the study
  Collection of serum IL-6 to identify a change from pre-post to analyze the effect protein isolates had on inflammation markers.
Normalized protein catabolic rate | Up to 12 weeks of the study
  Analysis of nPCR to identify a change from pre-post to analyze the effect protein isolates had on nPCR.

SECONDARY OUTCOMES:
Isoflavones - Serum values of Genistin and Daidzin | Up to 12 weeks of the study
  Collection of serum isoflavones (genistin and daidzin) to identify a change from pre-post to analyze the effect soy protein isolate had on inflammation markers that will be assessed via HPLC.
Uremic toxins - serum p-cresol sulfate and indoxyl sulfate | Up to 12 weeks of the study
  Collection of serum uremic toxins (p-cresol sulfate and indoxyl sulfate) to identify a change from pre-post to analyze the effect soy protein isolate had on inflammation markers that will be assessed via LC/MS.
Serum Amino acid profiles of essential and non-essential amino acids | Up to 12 weeks of the study
  Collection of serum amino acid profile of essential and non-essential amino acids to identify a change from pre-post to analyze the effect amino acids had on inflammation markers that will be assessed via LC/MS.
Malnutrition Inflammation Score | Up to 12 weeks of the study
  Assessment of malnutrition at baseline and post-intervention to determine nutritional status. There are a total of 10 questions that participants will answer. Scores are from as low as 0 to as high for 3 for each question. A score of 0 indicates normal whereas a score of 30 indicates severe malnutrition.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No